CLINICAL TRIAL: NCT02725788
Title: A Multi-Center, Prospective, Randomized Trial Comparing the Peripheral I.V. Catheter Complication Rates of Two Different Catheter Dressings
Brief Title: Trial Comparing Peripheral I.V. Catheter Complication Rates of Two Different Catheter Dressings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to futility
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM-05-013243
Record Dates: First submitted 2015-01-15; First posted 2016-04-01 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New PIV Dressing (Experimental): Bordered, notched dressing that covers, secures peripheral intravenous (PIV) catheter
  Interventions: Device: New PIV Dressing
- Standard PIV Dressing (Other): Film,adhesive dressing that covers, secures peripheral intravenous (PIV) catheter and used with a medical grade tape
  Interventions: Device: Standard PIV Dressing

INTERVENTIONS:
Device: New PIV Dressing — A commercially available breathable, transparent film dressing with a soft-cloth border, notch and securement tape strip. The dressing system is used in the study to cover a peripheral intravenous catheter insertion site and secure the catheter. Dressing system is to remain in place until the PIV catheter is discontinued which is anticipated to be 72 hours. The dressing and PIV site will be observed daily. If dressing excessively lifts from the skin, the dressing system will be replaced with the same, assigned dressing system. The number of dressing replacements and the duration of wear will be measured while the same study PIV catheter dwells, an average of 72 hours during the subject's hospitalization.
  Arms: New PIV Dressing
Device: Standard PIV Dressing — A commercially available breathable, transparent film dressing used with a one inch width piece of Transpore™ medical tape. The dressing system is used in the study to cover a peripheral intravenous catheter insertion site and secure the catheter. Dressing system is to remain in place until catheter is discontinued which is anticipated to be 72 hours. The dressing and PIV site will be observed daily. If dressing excessively lifts from the skin, the dressing system will be replaced with the same, assigned dressing system. The number of dressing replacements and the duration of wear will be measured while the same study PIV catheter dwells, an average of 72 hours during the subject's hospitalization.
  Arms: Standard PIV Dressing

SUMMARY:
A multi-center randomized control trial comparing the dressing wear times of two different transparent film dressings when used to secure peripheral intravenous catheters of hospitalized adult patients.

DETAILED DESCRIPTION:
A multi-center, prospective, randomized control trial comparing the dressing wear time, complication rates and cost of two different transparent film dressing when used as intended for peripheral intravenous catheter site protection and securement in five U.S. hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age, or of consenting age;
2. Admitted or going to be admitted to the hospital;
3. Requires peripheral IV therapy (catheter) for an anticipated 72 hours or longer;
4. Has an insertion site in the forearm or hand free of phlebitis, infiltration, dermatitis, burns, lesions or tattoos;
5. Demonstrates cooperation with a catheter insertion and the securement protocol; and
6. Patient or legally authorized representative is willing and able to provide written informed consent and authorization for use and disclosure of Protected Health Information

Exclusion Criteria:

1. Is a current participant or a past participant in this study;
2. If the subject already has a functioning PIV in place, not requiring a replacement catheter
3. If the study PIV catheter site will be placed below an old infusion site;
4. If the study PIV site needs to be immobilized with a splint or other device;
5. Has a documented or a known allergy or sensitivity to a medical adhesive product such as transparent film adhesive dressings, tapes, or liquid skin protectants;
6. Requires the application of a gauze pad, a topical ointment or solution under the dressing in addition to the prep(s) required in the protocol;
7. Will require a power injection through the study PIV catheter for a radiologic procedure during participation in this study;
8. Will require a numbing agent prior to PIV insertion; or
9. Will require the use of ultrasound for the PIV catheter insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Rupp, MD, Principal Investigator — University of Nebraska
Locations (5):
- United States (5):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of North Carolina, Chapel Hill, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Not required based on FDAA requirements

REFERENCES:
- [Background] Wood D. A comparative study of two securement techniques for short peripheral intravenous catheters. J Intraven Nurs. 1997 Nov-Dec;20(6):280-5. PMID 9423389
- [Background] Alexander M. Corrigan A. Infusion Nurses Society: Infusion nursing an evidence-based approach. St. Louis, Mo.: Saunders-Elsevier; 2010.
- [Background] Royer T. Improving short peripheral IV outcomes: a clinical trial of two securement methods. Journal of the Association for Vascular Access. 2003; 8(4): 45-49.
- [Background] Sheppard K, LeDesma M, Morris NL, O'Connor K. A prospective study of two intravenous catheter securement techniques in a skilled nursing facility. J Intraven Nurs. 1999 May-Jun;22(3):151-6. PMID 10640079
- [Background] Rosenthal K. Get a hold on costs and safety with securement devices. Nurs Manage. 2005 May;36(5):52-4. doi: 10.1097/00006247-200505000-00014. PMID 15879998
- [Background] Schears GJ. Summary of product trials for 10, 164 patients: comparing an intravenous stabilizing device to tape. J Infus Nurs. 2006 Jul-Aug;29(4):225-31. doi: 10.1097/00129804-200607000-00009. PMID 16858255
- [Background] Bausone-Gazda D, Lefaiver CA, Walters SA. A randomized controlled trial to compare the complications of 2 peripheral intravenous catheter-stabilization systems. J Infus Nurs. 2010 Nov-Dec;33(6):371-84. doi: 10.1097/NAN.0b013e3181f85be2. PMID 21079465
- [Background] Dunnett CW, Gent M. An alternative to the use of two-sided tests in clinical trials. Stat Med. 1996 Aug 30;15(16):1729-38. doi: 10.1002/(SICI)1097-0258(19960830)15:163.0.CO;2-M. PMID 8870155
- [Background] Hwang IK, Morikawa T. Design issues in noninferiority/equivalence trials. Drug Information journal 33: 1205-18, 1999.
- [Background] Tripathi S, Kaushik V, Singh V. Peripheral IVs: factors affecting complications and patency--a randomized controlled trial. J Infus Nurs. 2008 May-Jun;31(3):182-8. doi: 10.1097/01.NAN.0000317704.03415.b9. PMID 18496062
- [Background] Tripepi-Bova KA, Woods KD, Loach MC. A comparison of transparent polyurethane and dry gauze dressings for peripheral i.v. catheter sites: rates of phlebitis, infiltration, and dislodgment by patients. Am J Crit Care. 1997 Sep;6(5):377-81. PMID 9283675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 24, 2014 to May 12, 2015 at five U.S. hospitals
Groups:
- New Dressing: Bordered, notched film dressing sized to cover, secure peripheral venous (PIV) catheters
- Standard PIV Dressing: Film adhesive dressing used with medical grade tape and sized to cover, secure peripheral (PIV) catheters
Period: Overall Study
Arm/Group | New Dressing | Standard PIV Dressing
Started | 123 | 124
Completed | 122 | 122
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects randomized except 3 subjects who either failed to have the study dressing applied or whom the primary endpoint could not be ascertained
Groups:
- Total: Total of all reporting groups
Arm/Group | New Dressing | Standard PIV Dressing | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 78 | 155
  >=65 years | 45 | 44 | 89
Age, Continuous [Median (Full Range); unit: years] | 60 [18 to 93] | 60 [19 to 89] | 60 [18 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 118
  Male | 62 | 64 | 126
Region of Enrollment [Number; unit: participants]
  United States | 122 | 122 | 244
PIV catheter insertion location [Count of Participants; unit: Participants]
  Hand | 74 | 71 | 145
  Lower Forearm | 22 | 20 | 42
  Mid Forearm | 16 | 15 | 31
  Upper Forearm | 10 | 16 | 26

OUTCOME MEASURES:

1. Primary Outcome: Dressing Wear Time
Description: Dressing wear time is the time from dressing application to removal, i.e. catheter no longer needed or catheter-related complication occurs (remove dressing and catheter) OR excessive dressing lift requiring dressing replacement.
Time Frame: Dressing wear time was assessed daily and 8 month dressing wear data are presented
Population: All subjects randomized except three subjects who either failed to have a study dressing applied or whom could not have the primary endpoint ascertained.
Measure: Median (Full Range); unit: Days
Arm/Group | New Dressing | Standard PIV Dressing
Number analyzed (Participants) | 122 | 122
Days | 2.1 [0 to 7.0] | 2.1 [0 to 7.7]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | New Dressing | Standard PIV Dressing
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/124
Other Adverse Events (participants affected / at risk) | 0/123 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No